CLINICAL TRIAL: NCT02787746
Title: Safety and Efficacy of Donepezil in Mild to Moderate Alzheimer's Disease: A Multi-center Single-arm Study in China
Brief Title: Safety and Efficacy of Donepezil in Mild to Moderate Alzheimer's Disease
Acronym: STDMMAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Eisai China Inc. (Industry); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jianping Jia, Director of Neurology Department, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STD-CHINA-001
Record Dates: First submitted 2016-03-06; First posted 2016-06-01 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Disease
Keywords: AD; Donepezil; Safety
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: multi-center, single-arm, open labeling clinical trial
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- donepezil (Other): This is a multi-center single-arm study, which assess the safety and efficacy of donepezil in mild to moderate Alzheimer's disease in China.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Eligible patients were treated with Aricept® 10 mg/day for 20 weeks of study period. Aricept® should be taken at night, just prior to sleeping. If patient cannot endure 10mg/d，the dose could be reduce to 5mg/d for 4 weeks and then increase back to 10mg/d. Patients who could not endure the 10mg/d titration the 2nd time and were put back to 5mg/d or discontinuance of Aricept® should be considered as withdrawal from the study. There were a visit (visit 1) at week 0, the end of week 4 (visit 2) and the end of week 20 (visit 3), respectively.
  Other Names: Aricept

SUMMARY:
This study will evaluate the safety and Efficacy of donepezil in treatment of AD patients in China.

DETAILED DESCRIPTION:
This study is a multi-center, single-arm, open labeling clinical trial, which the objective is to evaluate the safety and Efficacy of donepezil in Alzheimer's disease( AD) patients in China, and investigate the relationship between Apo-E gene type with adverse events of donepezil.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 50 and 85 years of age.
2. Patients newly diagnosed as probable AD based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria and National Institute of Neurologic and Communicative Disorders and Stroke-AD and Related Disorders Association (NINCDS-ADRDA) criteria; Mild to moderate AD with Mini-Mental State Examination (MMSE) 10-24, modified Hachinski ischaemic scale (MHIS)≤4, Activity of daily life scale (ADL)≥23, and Hamilton Depression Scale (HAMD) <7.
3. MRI image supports the diagnosis of AD (medial temporal lobe atrophy, Fazekas scale of white matter lesions≤2 within 6 months prior to the screening).
4. 5mg daily of Donepezil for at least four weeks before the screening.
5. Patient with exclusive caregiver.
6. Patient should be ambulatory or ambulatory aided by a walker or cane.
7. With good eyesight and hearing, can cooperate with the examination and treatment.

Exclusion Criteria:

1. Patients with vascular dementia, other types of dementia or with other psychiatric or neurological disorders (e.g. delirium, depression, Parkinson's disease, etc.).
2. Patients with type I diabetes, obstructive lung disease or asthma, vitamin B12 or folic acid deficiency, thyroid dysfunction, severe liver or kidney dysfunction, severe cardiac insufficiency (congestive heart failure, myocardial infarction, sick sinus syndrome, II-III degree atrioventricular block or heart rate<50 beats/minute [bpm]).
3. Epilepsy or head trauma resulting in unconsciousness that occurred in the two years prior to the screening.
4. Patients with hematologic diseases (such as anemia, granulocytes, leukemia, etc.), tumor, neoplasms within 2 years prior to the screening.
5. Patients with a history of alcohol dependence and drug abuse.
6. Patients with known hypersensitivity to medicines or foods;
7. Patients taking anticholinergic agents or antihistaminic agents;
8. Patients who had been hospitalized continuously for more than 3 months before the screening.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cuibai Wei, MD,PhD, Study Director — Dept of Neurology, Beijing Friendship Hospital, Capital Medical University
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
No data will be share.

REFERENCES:
- [Derived] Jia J, Wei C, Chen W, Jia L, Zhou A, Wang F, Tang Y, Xu L. Safety and Efficacy of Donepezil 10 mg/day in Patients with Mild to Moderate Alzheimer's Disease. J Alzheimers Dis. 2020;74(1):199-211. doi: 10.3233/JAD-190940. PMID 31985467

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: Each enrolled patient received donepezil 10 mg/day (Aricept, two 5 mg-pills, Eisai China Inc, SuZhou, China) every night before sleeping for 20 weeks. If a patient could not tolerate 10 mg/day, the dosage for the patient could be reduced to 5 mg/day for 4 weeks and then increased back to 10 mg/day. If this patient still could not tolerate the 10 mg/day dosage and returned back to 5 mg/day or discontinued the donepezil treatment, he/she should be deemed to have quit the study.
Period: Overall Study
Arm/Group | Donepezil
Started | 241
Completed | 93
Not Completed | 148
Not completed — Adverse Event | 42
Not completed — Withdrawal by Subject | 65
Not completed — Failure to up-titrate to 10mg/day: 12 patients; Other reasons: 30 patients | 41

BASELINE CHARACTERISTICS:
Groups:
- Donepezil: Daily single dose of donepezil 10mg
Arm/Group | Donepezil
Number analyzed (Participants) | 241
Age, Customized [Count of Participants; unit: Participants]
  <65 Years old | 44
  65-74 Years old | 84
  75-84 Years old | 110
  ≥85 Years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Count of Participants; unit: Participants]
  ≤55 kg | 97
  56-65 kg | 74
  66-75 kg | 47
  >75 kg | 23
Heart rate [Mean (Standard Deviation); unit: beat/min] | 72.35 (9.49)
Corrected QT interval (QTc) [Mean (Standard Deviation); unit: msec] | 419.16 (29.9)
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] | 23.16 (14.09)
Past Medical history [Count of Participants; unit: Participants]
  Cardiovascular diseases | 39
  Neurologic disease | 58
  Mental disease | 10
  Liver disease | 13
  Gastrointestinal diseases | 17
  Other disease | 46
  No disease | 58
Concomitant drugs [Count of Participants; unit: Participants]
  Cardiovascular drugs | 22
  Central nervous system drugs | 106
  Antipsychiatric drugs | 18
  Hepatology drugs | 1
  Gastrointestinal diseases drugs | 5
  Other drugs | 3
  Did not use | 86
MMSE [Mean (Standard Deviation); unit: score] — MMSE,Mini-Mental State Examination (range 0-30). A higher score indicates better cognitive function.
  score | 18.69 (4.35)
ADCS-ADL(Alzheimer's disease cooperative study - activities of daily living) [Mean (Standard Deviation); unit: Score unit] — ADCS-ADL (Alzheimer's disease cooperative study - activities of daily living) score (range 0 to 78), a higher score indicates better ADL function)
  Score unit | 53.29 (11.55)
HAMD [Mean (Standard Deviation); unit: Score unit] — HAMD, Hamilton Depression Scale (score range 0 to 52). A score >7and ≤17 indicates mild depression; a score >17 and ≤24 indicates moderate depression; and a score >24 indicates severe depression.
  Score unit | 3.09 (2.56)
Previous duration of donepezil 5mg/d therapy [Mean (Standard Deviation); unit: day] | 70.97 (123.95)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: Physical examinations such as vital signs and weight, clinical laboratory tests, and electrocardiograms (ECGs) during the 20 weeks.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 241
Participants | 93

2. Secondary Outcome: Number of Patients Who Withdrew From the Trial Due to Adverse Events.
Description: Number of patients who withdrew due to adverse events
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 241
Participants | 42

3. Secondary Outcome: Changes in Mini-Mental State Examination Scores From Baseline
Description: Comparison of Mental state examination (MMSE) scores (range 0-30) at 4 weeks and 20 weeks with baseline in mild to moderate AD patients. A higher score indicates better cognitive function.Higher score indicates better cognition function.
Time Frame: Baseline, 4, 20 weeks
Population: 241 patients were included in the full analysis set (FAS) and 93 patients who completed the study constituted the per-protocol set (PPS). Therefore, FAS last-observation-carried-forward [LOCF] and PPS [LOCF] included 241 and 93 patients, respectively.
  FAS [actual data] at baseline, Week 4 and Week 20 included 238, 145 and 94 patients, respectively.
  PPS [actual data] at baseline, Week 4 and Week 20 included 148, 113 and 93 patients, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; Week 4; Change From Baseline at Week 4; Week 20; Change From Baseline at Week 20: Daily single dose of donepezil 10mg
Arm/Group | Baseline | Week 4 | Change From Baseline at Week 4 | Week 20 | Change From Baseline at Week 20
Number analyzed (Participants) | 241 | 241 | 241 | 241 | 241
score on a scale
  FAS LOCF | 18.69 (4.35) | 19.12 (5.06) | 0.44 (2.51) | 19.07 (5.30) | 0.39 (2.64)
  FAS (actual data): number analyzed (Participants) | 238 | 145 | 145 | 94 | 94
  FAS (actual data) | 18.69 (4.35) | 18.87 (5.76) | 0.72 (3.19) | 19.62 (5.8) | 0.97 (3.18)
  PPS LOCF: number analyzed (Participants) | 93 | 93 | 93 | 93 | 93
  PPS LOCF | 18.45 (4.39) | 19.22 (5.18) | 0.77 (2.53) | 19.11 (5.54) | 0.66 (2.74)
  PPS (actual data): number analyzed (Participants) | 148 | 113 | 113 | 93 | 93
  PPS (actual data) | 18.45 (4.39) | 19.33 (5.53) | 1.01 (2.86) | 19.57 (5.81) | 0.94 (3.18)

4. Secondary Outcome: Changes in Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Scores From Baseline
Description: Comparison of Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) scores (range 0-78) at 4 weeks and 20 weeks with baseline scores in patients with mild to moderate Alzheimer's Disease. A higher score indicates better activities of daily living (ADL).
Time Frame: Baseline, 4, 20 weeks
Population: 241 patients were included in the FAS and 93 patients who completed the study constituted the PPS. Therefore, FAS [LOCF] and PPS [LOCF] included 241 and 93 patients, respectively.
  FAS [actual data] at baseline, Week 4 and Week 20 all included 42 patients, while PPS [actual data] at baseline, Week 4 and Week 20 all included 26 patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Week 4 | Change From Baseline at Week 4 | Week 20 | Change From Baseline at Week 20
Number analyzed (Participants) | 241 | 241 | 241 | 241 | 241
score on a scale
  FAS LOCF | 53.29 (11.55) | 53.71 (12.97) | 0.43 (7.34) | 53.62 (12.82) | 0.33 (7.47)
  FAS (actual data): number analyzed (Participants) | 42 | 42 | 42 | 42 | 42
  FAS (actual data) | 34.76 (14.04) | 33.31 (13.75) | -0.66 (6.04) | 30.86 (11.01) | -1.15 (11.04)
  PPS LOCF: number analyzed (Participants) | 93 | 93 | 93 | 93 | 93
  PPS LOCF | 54.31 (10.63) | 54.35 (12.50) | 0.04 (6.20) | 54.19 (12.25) | -0.12 (6.44)
  PPS (actual data): number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
  PPS (actual data) | 33.31 (13.58) | 32.71 (13.5) | -0.65 (6.69) | 30.9 (11.07) | -1.13 (11.11)

5. Secondary Outcome: Correlation Between Apolipoprotein E.(APOE) Genotype and Incidence of Adverse Events of Donepezil
Description: Comparison of incidence of adverse events among patients with different APOE genotypes
Time Frame: 20 weeks
Population: 115 patients in the safety set had their APOE gene sequenced and have data on their APOE genotype. Among these patients, 1 carries APOE ɛ2/ɛ2, 58 carry APOE ɛ3/ɛ3, 7 carry APOE ɛ4/ɛ4, 11 carry APOE ɛ2/ɛ3, 1 carries APOE ɛ2/ɛ4, and 37 carry APOE ɛ3/e4.
Measure: Count of Participants; unit: Participants
Groups:
- APOE ɛ2/ɛ2 Carriers: Number of APOE ɛ2/ɛ2 carriers
- APOE ɛ3/ɛ3 Carriers: Number of APOE ɛ3/ ɛ3 carriers
- APOE ɛ4/ɛ4 Carriers: Number of APOE ɛ4/ɛ4 carriers
- APOE ɛ2/ɛ3 Carriers: Number of APOE ɛ2/ɛ3 carriers
- APOE ɛ2/ɛ4 Carriers: Number of APOE ɛ2/ɛ4 carriers
- APOE ɛ3/e4 Carriers: Number of APOE ɛ3/e4 carriers
Arm/Group | APOE ɛ2/ɛ2 Carriers | APOE ɛ3/ɛ3 Carriers | APOE ɛ4/ɛ4 Carriers | APOE ɛ2/ɛ3 Carriers | APOE ɛ2/ɛ4 Carriers | APOE ɛ3/e4 Carriers
Number analyzed (Participants) | 1 | 58 | 7 | 11 | 1 | 37
Participants
  Numbe of patients who experienced adverse events | 0 | 34 | 5 | 6 | 0 | 13
  Number of patients who did not experience adverse events | 1 | 24 | 2 | 5 | 1 | 24
Statistical Analysis 1: Comparison: APOE ɛ2/ɛ2 Carriers; Age (>75y vs ≤75y）; Test type: Other; p = 0.9744, Regression, Logistic; Odds Ratio (OR) = 0.988, 95% CI 2-sided [0.466 to 2.095]
Statistical Analysis 2: Comparison: APOE ɛ2/ɛ2 Carriers; APOE ɛ4 (carrier vs non-carrier); Test type: Other; p = 0.3288, Regression, Logistic; Odds Ratio (OR) = 3.420, 95% CI 2-sided [0.290 to 40.354]
Statistical Analysis 3: Comparison: APOE ɛ2/ɛ2 Carriers; Concomitant medication：Gastrointestinal drugs; Test type: Other; p = 0.5732, Regression, Logistic; Odds Ratio (OR) = 2.107, 95% CI 2-sided [0.158 to 28.171]
Statistical Analysis 4: Comparison: APOE ɛ2/ɛ2 Carriers; Concomitant medication：Hypoglycemic drugs; Test type: Other; p = 0.9694, Regression, Logistic; Odds Ratio (OR) = 0.976, 95% CI 2-sided [0.281 to 3.387]
Statistical Analysis 5: Comparison: APOE ɛ2/ɛ2 Carriers; Concomitant medication：Cardiovascular and Cerebrovascular drugs; Test type: Other; p = 0.0396, Regression, Logistic; Odds Ratio (OR) = 2.221, 95% CI 2-sided [1.039 to 4.748]
Statistical Analysis 6: Comparison: APOE ɛ2/ɛ2 Carriers; Concomitant medication：Hepatology drugs; Test type: Other; p = 0.5889, Regression, Logistic; Odds Ratio (OR) = 2.056, 95% CI 2-sided [0.151 to 28.074]
Statistical Analysis 7: Comparison: APOE ɛ2/ɛ2 Carriers; Duration of previous donepezil 5mg/d therapy (day); Test type: Other; p = 0.1181, Regression, Logistic; Odds Ratio (OR) = 1.004, 95% CI 2-sided [0.999 to 1.008]

6. Secondary Outcome: APOE Genotype
Description: A patient's APOE genotype (ɛ2/ɛ2, ɛ3/ɛ3, ɛ4/ɛ4, ɛ2/ɛ3, ɛ2/ɛ4 and ɛ3/e4) was tested by tested by Sanger sequencing from blood collected from the the patient at Visit 2.
  APOE genotype is not mandatory
Time Frame: 4 weeks
Population: 115 patients in the study had their APOE genotype tested by Sanger sequencing from blood collected from the the patient at Visit 2.
Measure: Count of Participants; unit: Participants
Groups:
- Donepezil: Each patient took daily single dose of donepezil 10mg
Arm/Group | Donepezil
Number analyzed (Participants) | 115
Participants
  APOE ɛ2/ɛ2 | 1
  APOE ɛ3/ɛ3 | 58
  APOE ɛ4/ɛ4 | 7
  APOE ɛ2/ɛ3 | 11
  APOE ɛ2/ɛ4 | 1
  APOE ɛ3/e4 | 37

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | Donepezil
All-Cause Mortality (participants affected / at risk) | 0/241
Serious Adverse Events (participants affected / at risk) | 3/241
Other Adverse Events (participants affected / at risk) | 93/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=241)
Emesis (Gastrointestinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=241)
anemia (Blood and lymphatic system disorders) | 1 (1)
Hyperhomocysteinemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiac discomfort (Cardiac disorders) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 1 (1)
hypogastralgia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Gastritis (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 8 (8)
hygrostomia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
fever (General disorders) | 1 (1)
abnormal liver function (Hepatobiliary disorders) | 2 (2)
urocystitis (Infections and infestations) | 1 (1)
shingles (Infections and infestations) | 2 (2)
upper respiratory infection (Infections and infestations) | 2 (2)
urinary tract infection (Infections and infestations) | 5 (5)
bacterial infection (Infections and infestations) | 1 (1)
pulmonary infection (Infections and infestations) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 1 (1)
thoracic injury (Injury, poisoning and procedural complications) | 1 (1)
Elevated alanine aminotransferase (Investigations) | 1 (1)
Decreased aspartate aminotransferase (Investigations) | 1 (1)
Decreased blood albumin (Investigations) | 1 (4)
Elevated blood bilirubin (Investigations) | 2 (2)
Reduced blood chloride (Investigations) | 2 (2)
Increased blood creatine phosphokinase (Investigations) | 2 (2)
Increased blood creatinine (Investigations) | 3 (3)
Increased blood glucose (Investigations) | 2 (2)
Decreased blood lactate dehydrogenase (Investigations) | 1 (1)
Increased blood lactate dehydrogenase (Investigations) | 1 (1)
Decreased blood sodium (Investigations) | 2 (2)
Increased blood urea (Investigations) | 2 (2)
Abnormal ECG (Investigations) | 4 (4)
Abnormal EEG (Investigations) | 1 (1)
Reduced heart rate (Investigations) | 3 (4)
Decreased red blood cell count (Investigations) | 1 (1)
Urinary erythrocyte positive (Investigations) | 1 (1)
Increased white blood cell count (Investigations) | 1 (1)
Urine leukocyte positive (Investigations) | 3 (3)
Increased platelet count (Investigations) | 1 (1)
Decreased blood alkaline phosphatase (Investigations) | 1 (1)
Decreased blood creatine phosphokinase (Investigations) | 1 (1)
diabetes (Metabolism and nutrition disorders) | 2 (2)
hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Loss of appetite (Metabolism and nutrition disorders) | 3 (3)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes (Metabolism and nutrition disorders) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 5 (5)
Skeletal muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Physical discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (Nervous system disorders) | 4 (5)
Memory impairment (Nervous system disorders) | 1 (1)
Drowsiness (Nervous system disorders) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 2 (2)
sleep disorder (Psychiatric disorders) | 5 (6)
Amnesia (Psychiatric disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
hidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
skin disease (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-10-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT02787746/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02787746/SAP_001.pdf
  • Informed Consent Form (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02787746/ICF_002.pdf